CLINICAL TRIAL: NCT03727854
Title: Effect of Premeal Consumption of Protein-enriched, Dietary Fiber-fortified Cereal Bar on Long-term Glycemic Control in Patients With Type 2 Diabetes
Brief Title: Effect of Premeal Protein-bar on Glycemic Control in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young Min Cho, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-1804-120-940
Record Dates: First submitted 2018-10-31; First posted 2018-11-01 (Actual); Results first posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Patients With Type 2 Diabetes
Keywords: protein-enriched bar; glycemic control; type 2 diabetes; long term
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Premeal protein group (Experimental): Premeal protein enriched bar with dietary modification
  Interventions: Dietary Supplement: Premeal protein enriched bar; Behavioral: Dietary modification
- Dietary modofication only group (Other): Dietary modification only
  Interventions: Behavioral: Dietary modification

INTERVENTIONS:
Dietary Supplement: Premeal protein enriched bar — Subjects in the intervention group will intake protein enriched bar 15 minutes before each meals (at least twice a day).
  Arms: Premeal protein group
Behavioral: Dietary modification — Subjects in this group will follow diabetes diet education.

SUMMARY:
The aim of this study is to evaluate the effect of premeal protein-enriched bar in long-term glycemic control in patients with type 2 diabetes mellitus. Glucose levels in subjects who intake premeal protein-enriched bar with dietary modification will be compared to those in subjects who only do the dietary modification.

DETAILED DESCRIPTION:
Forty subjects with type 2 diabetes will be recruited. Every subject will be randomized in two groups, which are premeal protein bar with dietary modification group and dietary modification only group. The study will be conducted for 12 weeks for each participants. All participants will receive diabetes diet education. Intervention group will consume protein-enriched bar before each meals (at least twice a day) and control group will follow diabetes diet education without other additional supplements. Primary outcome is change of HbA1c from baseline for 12 weeks, and secondary outcomes are changes of fasting blood glucose level, body weight, waist circumference, blood lipid level, HOMA-IR and HOMA-beta from baseline for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5~35 kg/m2
* Type 2 diabetes patients
* Fasting blood glucose ≥ 126 mg/dl or
* HbA1c ≥ 6.5% or
* Subjects who were previously diagnosed with type 2 diabetes and who have been treated with lifestyle modification only, oral anti-diabetic drugs or basal insulin.

Exclusion Criteria:

* HbA1c < 6.5% or > 10%
* Subjects using insulin other than basal insulin
* Subjects who have newly started or have changed anti diabetic drugs within 3 months
* Subjects who are allergic to grains, nuts, legumes and milk
* Previous history of gastrointestinal surgery (except for hemorrhoid surgery, appendectomy surgery and hernia surgery)
* Subjects with chronic unstable disease
* Subjects with cognitive impairments who are not able to follow the study protocol
* Females who are pregnant or doing breast feeding
* Subjects with Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels of higher than 3 times of upper normal ranges
* Subjects with hemoglobin level of less than 10.0 g/dL
* Subjects with alcohol addiction or drug abuse

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Group1: Premeal protein enriched bar with dietary modification
  Premeal protein enriched bar: Subjects in the intervention group will intake protein enriched bar 15 minutes before each meals (at least twice a day).
  Dietary modification: Subjects in this group will follow diabetes diet education.
- Group2: Dietary modification only
  Dietary modification: Subjects in this group will follow diabetes diet education.
Period: Overall Study
Arm/Group | Group1 | Group2
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group1 | Group2 | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (5.2) | 64.1 (8.3) | 64.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline
Time Frame: 0 week, 12 weeks
Measure: Mean (Standard Deviation); unit: % (HbA1c)
Arm/Group | Group1 | Group2
Number analyzed (Participants) | 20 | 20
% (HbA1c) | 0.015 (0.706) | 0.030 (0.354)
Statistical Analysis 1: Comparison: Group1 vs Group2; Test type: Superiority; p = 0.933, t-test, 2 sided

2. Secondary Outcome: Change in Fasting Blood Glucose Level From Baseline
Time Frame: 0 week, 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group1 | Group2
Number analyzed (Participants) | 20 | 20
mg/dL | 1.9 (26.2) | 1.6 (25.5)
Statistical Analysis 1: Comparison: Group1 vs Group2; Test type: Superiority; p = 0.971, t-test, 2 sided

3. Secondary Outcome: Change in Body Weight From Baseline
Time Frame: 0 week, 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Group1 | Group2
Number analyzed (Participants) | 20 | 20
kg | 0.21 (0.98) | 0.03 (1.26)
Statistical Analysis 1: Comparison: Group1 vs Group2; Test type: Superiority; p = 0.608, t-test, 2 sided

4. Secondary Outcome: Change in Waist Circumference From Baseline
Time Frame: 0 week, 12 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Group1 | Group2
Number analyzed (Participants) | 20 | 20
cm | 0.70 (3.73) | 0.15 (3.15)
Statistical Analysis 1: Comparison: Group1 vs Group2; Test type: Superiority; p = 0.617, t-test, 2 sided

5. Secondary Outcome: Change in Blood Triglyceride Level From Baseline
Time Frame: 0 week, 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group1 | Group2
Number analyzed (Participants) | 20 | 20
mg/dL | -5.05 (50.74) | -1.30 (54.21)
Statistical Analysis 1: Comparison: Group1 vs Group2; Test type: Superiority; p = 0.823, t-test, 2 sided

6. Secondary Outcome: Change in Blood High-density Lipoprotein Level From Baseline
Time Frame: 0 week, 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group1 | Group2
Number analyzed (Participants) | 20 | 20
mg/dL | -3.70 (6.38) | -5.05 (16.91)
Statistical Analysis 1: Comparison: Group1 vs Group2; Test type: Superiority; p = 0.740, t-test, 2 sided

7. Secondary Outcome: Change in Blood Low-density Lipoprotein Level From Baseline
Time Frame: 0 week, 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group1 | Group2
Number analyzed (Participants) | 20 | 20
mg/dL | 2.90 (17.31) | -0.70 (20.44)
Statistical Analysis 1: Comparison: Group1 vs Group2; Test type: Superiority; p = 0.551, t-test, 2 sided

8. Secondary Outcome: Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) From Baseline
Description: Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) is an index to estimate the insulin resistance of a subject. HOMA-IR is defined as ( glucose (mg/dl) X insulin (uIU/ml) ) / 405.
Time Frame: 0 week, 12 weeks
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Group1 | Group2
Number analyzed (Participants) | 20 | 20
units | -1.00 (5.11) | -0.46 (1.67)
Statistical Analysis 1: Comparison: Group1 vs Group2; Test type: Superiority; p = 0.652, t-test, 2 sided

9. Secondary Outcome: Change in Homeostatic Model Assessment of β-cell Function (HOMA-beta) From Baseline
Description: as for outcome 8
Time Frame: 0 week, 12 weeks
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Group1 | Group2
Number analyzed (Participants) | 20 | 20
units | -35.53 (196.36) | -13.9 (58.40)
Statistical Analysis 1: Comparison: Group1 vs Group2; Test type: Superiority; p = 0.639, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Group1 | Group2
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT03727854/Prot_SAP_000.pdf